CLINICAL TRIAL: NCT00851552
Title: A Phase II Study of VDR (VELCADE™, DOXIL® and RITUXAN™) in Relapsed/Refractory Diffuse Large B-cell Lymphoma
Brief Title: Bortezomib, Doxorubicin Hydrochloride Liposome, and Rituximab in Treating Patients With Diffuse Large B-Cell Lymphoma That Has Relapsed or Not Responded to Treatment
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of sponsor support
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Ortho Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000635486; RPCI-I-136508
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Results first posted 2014-07-21 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-06

CONDITIONS: Lymphoma
Keywords: recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; anaplastic large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Large-Cell, Anaplastic | interventions — Rituximab; Bortezomib; Gene Expression Profiling; Polymerase Chain Reaction; Amplified Fragment Length Polymorphism Analysis; Flow Cytometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: rituximab — Given IV
Drug: bortezomib — Given IV
Drug: pegylated liposomal doxorubicin hydrochloride — Given IV
Genetic: gene expression analysis — Correlative Study
Genetic: polymerase chain reaction — Correlative Study
Genetic: polymorphism analysis — Correlative Study
Genetic: proteomic profiling — Correlative Study
Other: flow cytometry — Correlative Study
Other: laboratory biomarker analysis — Correlative Study

SUMMARY:
RATIONALE: Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the cancer. Drugs used in chemotherapy, such as doxorubicin hydrochloride liposome, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as rituximab, can block cancer cell growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cell-killing substances to them. Giving bortezomib together with doxorubicin hydrochloride liposome and rituximab may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving bortezomib together with doxorubicin hydrochloride liposome and rituximab works in treating patients with diffuse large B-Cell lymphoma that has relapsed or not responded to treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the overall objective response rate (i.e., complete and partial response) in patients with relapsed or refractory, CD20-positive, diffuse large B-cell lymphoma treated with bortezomib, pegylated liposomal doxorubicin hydrochloride, and rituximab.

Secondary

* To assess the toxicity/safety profile associated with this regimen.
* To conduct correlative translational research studies.

OUTLINE: Patients receive bortezomib IV on days 1, 4, 8, and 11, pegylated liposomal doxorubicin hydrochloride IV on day 11, and rituximab IV on day 8. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.

Tissue and blood samples are collected periodically for correlative studies. Samples are analyzed for expression of CD11b/CD18, CD32, CD 33, CD62, CD64, CD69, and CD56 by flow cytometric analysis of neutrophils, NK cells, and monocytes; antibody-dependent cellular and complement-mediated cytotoxicity; and genotypic analysis of polymorphisms by PCR. Autologous neoplastic B-cells derived from tissue samples are used for genetic and protein profiling.

After completion of study therapy, patients are followed periodically for 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of CD20-positive diffuse large B-cell lymphoma, including any of the following morphological variants:

  * Centroblastic
  * Immunoblastic
  * T-cell/histiocyte-rich
  * Anaplastic
  * Mediastinal (thymic) large B-cell lymphoma
  * Intravascular large B-cell lymphoma
* Relapsed or refractory disease
* Measurable disease, defined as tumor size 2 cm²
* Must have received ≥ 1 prior standard chemotherapy regimen
* No Burkitt or precursor B-lymphoblastic lymphoma
* No brain involvement or evidence of CNS lymphoma

PATIENT CHARACTERISTICS:

* Karnofsky performance status (PS) 70-100% OR ECOG PS 0-2
* Life expectancy ≥ 12 weeks
* Absolute neutrophil count ≥ 1,500/μL*
* Platelet count ≥ 100,000/μL*
* Creatinine < 2.5 mg/dL OR > 40 mL/min*
* Hemoglobin > 8.0 g/dL*
* AST/ALT < 2 times upper limit of normal (ULN) (< 3 times ULN with liver involvement)*
* Alkaline phosphatase < 2 times ULN (< 3 times ULN with liver involvement)*
* Total bilirubin < 2 times ULN (< 3 times ULN with liver involvement or Gilbert disease)* NOTE: *Unless attributable to non-Hodgkin lymphoma
* LVEF ≥ 50% by MUGA scan or ECHO
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after completion of therapy
* No HIV positivity
* No hepatitis B positivity
* Peripheral neuropathy < grade 2 as defined by NCI CTCAE v 3.0
* No history of uncontrolled orthostatic hypotension
* None of the following cardiac conditions:

  * Myocardial infarction within the past 6 months
  * New York Heart Association class II-IV congestive heart failure
  * Uncontrolled angina
  * Severe uncontrolled ventricular arrhythmias
  * Clinically significant pericardial disease
  * ECG evidence of acute ischemic or active conduction system abnormalities
* No hypersensitivity to bortezomib, boron, or mannitol
* No history of allergic reactions to compounds containing boron, mannitol, bortezomib, conventional formulation of doxorubicin hydrochloride, or the components of pegylated liposomal doxorubicin hydrochloride
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Poorly controlled hypertension
  * Diabetes mellitus
  * Serious medical or psychiatric conditions that would interfere with adherence to or completion of this study
* No other primary malignancy except squamous cell or basal cell carcinoma of the skin, in situ carcinoma of the cervix, superficial bladder carcinoma, or previously treated localized prostate cancer with normal PSA levels and disease-free for ≥ 5 years

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from significant toxicity associated with prior surgery, radiotherapy, chemotherapy, or immunotherapy
* Prior rituximab or other monoclonal immunotherapy allowed
* More than 4 weeks since prior investigational drugs
* More than 4 weeks since prior chemotherapy
* More than 4 weeks since prior major surgery, other than diagnostic surgery
* No prior doxorubicin hydrochloride (or equivalent) anthracycline treatment exceeding 400 mg/m²
* No concurrent corticosteroids, except to control a transient inflammatory reaction (i.e., skin rash or hives)

  * Concurrent non-steroidal hormones administered for non-lymphoma related conditions (e.g., insulin for diabetes) allowed
* No concurrent radiotherapy
* No other concurrent antitumor or chemotherapeutic agents
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Myron S. Czuczman, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- VDR: Velcade, Doxil, and Rituxan: VELCADE - 1.3mg/m2 IV, days 1, 4, 8, 11 every 21 days x 6 cycles DOXIL - 30 mg/m2 IV, day 11 every 21 days x 6 cycles RITUXAN - 375 mg/m2 IV, day 8 every 21 days x 6 cycles
Period: Overall Study
Arm/Group | VDR: Velcade, Doxil, and Rituxan
Started | 9
Completed | 2
Not Completed | 7
Not completed — Death | 2
Not completed — Adverse Event | 1
Not completed — Disease Progression | 4

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Arm/Group | VDR: Velcade, Doxil, and Rituxan
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.78 (18.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Antitumor Efficacy in Terms of Overall, Complete, and Partial Response Rates and Time to Progression at Weeks 9 and 21
Time Frame: at weeks 9 and 21
Population: Due to the study's early termination and inadequate number of patients, no patients were analyzed.
Arm/Group | VDR: Velcade, Doxil, and Rituxan
Number analyzed (Participants) | 0

2. Secondary Outcome: Safety
Time Frame: 2 years
Population: Due to the study's early termination and inadequate number of patients, no patients were analyzed.
Arm/Group | VDR: Velcade, Doxil, and Rituxan
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | VDR: Velcade, Doxil, and Rituxan
Serious Adverse Events (participants affected / at risk) | 5/9
Other Adverse Events (participants affected / at risk) | 7/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VDR: Velcade, Doxil, and Rituxan (N=9)
Myocardial infarction (Cardiac disorders) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 2 (2)
Troponin I increased (Investigations) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VDR: Velcade, Doxil, and Rituxan (N=9)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Platelet disorder (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (10)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (5)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3)
Chills (General disorders) | 2 (2)
Fatigue (General disorders) | 1 (2)
Pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Cytokine release syndrome (Immune system disorders) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Troponin increased (Investigations) | 1 (1)
Weight decreased (Investigations) | 1 (3)
Anorexia (Metabolism and nutrition disorders) | 1 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 2 (2)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to the study's early termination and inadequate number of patients, no patients were analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes